CLINICAL TRIAL: NCT04125628
Title: Effects of Head and Neck Cooling on Functional Ability and Fatigue of Multiple Sclerosis
Brief Title: Exercise on Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 5. Multiple Sclerosis
Record Dates: First submitted 2019-10-08; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: Uthoff's phenomenon; Thermosensitivity; Functional capacity; Exercise intolerance
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with cooling (Experimental): Assigned Interventions 10 MS patients (aged 25----50 years) with Expanded Disability Status Scale between 2 to 6.5 have agreed to participate in this study. The exercise training session involved head cooling and neck wraps. The exercise training session consisted of 40 min continuous cycling where the participants performed an incremental sub-maximal exercise protocol beginning at 45 W, increasing 10 W every 10 min for a total of four stages on a semirecumbent cycle ergometer in a 20oC room. Before and after the completion of the session each participant performed a variety of functional ability tests. The evaluation of the core temperature and the assessment of the patient's quality of life also was performed.
  Interventions: Behavioral: Exercise with cooling
- Exercise without cooling (Active Comparator): 10 MS patients (aged 25----50 years) with Expanded Disability Status Scale between 2 to 6.5 have agreed to participate in this study. The exercise session performed without cooling. The exercise training session consisted of 40 min continuous cycling where the participants performed an incremental sub-maximal exercise protocol beginning at 45 W, increasing 10 W every 10 min for a total of four stages on a semirecumbent cycle ergometer in a 20oC room. Before and after the completion of the session each participant performed a variety of functional ability tests. The evaluation of the core temperature and the assessment of the patient's quality of life also was performed.
  Interventions: Behavioral: Exercise without cooling

INTERVENTIONS:
Behavioral: Exercise with cooling — The exercise training session involved head cooling and neck wraps. Participants followed a 40-minute continuous cycling where they performed an incremental sub-maximal exercise protocol beginning at 45 W, increasing 10 W every 10 min for a total of four stages on a semirecumbent cycle ergometer in a 20oC room. Before and after the completion of the condition each participant performed a variety of functional ability tests. The evaluation of the core temperature and the assessment of the patient's quality of life also was performed
  Arms: Exercise with cooling
Behavioral: Exercise without cooling — The exercise session performed without cooling. Participants followed a 40-minute continuous cycling where they performed an incremental sub-maximal exercise protocol beginning at 45 W, increasing 10 W every 10 min for a total of four stages on a semirecumbent cycle ergometer in a 20oC room. Before and after the completion of the session each participant performed a variety of functional ability tests. The evaluation of the core temperature and the assessment of the patient's quality of life also was performed.
  Arms: Exercise without cooling

SUMMARY:
Multiple sclerosis (MS) patients are characterized by thermoregulatory failure, known as Uthoff's phenomenon. Precisely, 60-80% of the MS patients present adverse clinical symptoms when their body temperature is increased. Thus, the development of treatment strategies to overcome the thermoregulatory problem in these patients is crucial. Given that cooling has been proposed as an effective method, the aim of this study was to examine whether the application of head cooling therapy during an exercise training session is capable to prevent the core temperature increase and to improve the patient's functional ability and quality of life.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) mostly affects young individuals aged between 20 to 40 years and is the leading cause of morbidity and disability in young. Most of the MS patients experience motor symptoms such as ataxia, tremor, dizziness, limb weakness and vertigo that induce gait difficulty. More precisely, it has been reported that in around 85% of patients diagnosed with MS the gait difficulties are the main problem, which increases the risk for falls. Except for the motor difficulties, MS patients experience multiple physical, cognitive and neurological symptoms that reduce their quality of life. Also, fatigue is another frequent symptom, which is considered among the most disabling symptoms. MS patients 10 years after the onset of the disease become unable to perform housekeeping and employment responsibilities, and as a consequence, the patients experience high depression rates while the suicide incidence is high, varying from 28.6% to 2.5% in these patients. Over the past 15 years a variety of studies have proved that exercise training in patients with chronic diseases, improve their functional capacity and quality of life, and accordingly are capable of performing their daily living activities independently, while it can reduce depression and delay the progression of the disease's symptoms. Nevertheless, MS patients for many years were advised not to participate in exercise training programs because there was a perception that exercise could worsen the disease symptoms due to increased body temperature. Indeed 60-80% of the MS patients present adverse clinical symptoms when their body temperature is increased not only due to physical working but even when immersing in hot water or by exposure to infrared lamps or the sun. Since MS has a severe economic impact as it affects mostly young adults in their most productive years and leads to loss of work capacity and exercise training has the potential to prevent or ameliorate this loss, the need to develop new treatment strategies that could overcome the thermoregulatory problem during exercise is crucial. Therefore, it has been proposed that active precooling is considered an effective treatment for reducing the consequences of induced-heat stress due to exercise. Therefore, this study will examine whether a session of pre-cooling could improve the functional ability of patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (no menses for the last year at least);
* Osteoporosis patients (female): T-score<-2.5 at the femoral neck (or other anatomical site);
* Osteoporosis patients (male): T-score<-2.5 at the femoral neck (or other anatomical site)
* Osteopenia patients (female): T-score<-1.0 at the femoral neck (or other anatomical site);
* Osteopenia patients (male): T-score<-1.0 at the femoral neck (or other anatomical site)
* Patients taking drugs/ supplements for osteoporosis will be accepted in the study after going through a wash-up period

Exclusion Criteria:

* Women with irregular menses (i.e. with no established menopause)
* Patients taking medications for other diseases known to interfere with bone metabolism
* Patients with other chronic diseases (e.g. diabetes)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Core Temperature | Change from baseline to after 40 minutes of continous cycling.
  The core temperature was measured using a telemetric capsule or (e-Celsius Performance, BodyCap, Caen, France). Temperature at the skin surface was recorded every second at four sites using iBUTTON sensors (type DS1921 H, Maxim/Dallas Semiconductor Corp., USA) [Tsk; 0.3 (chest C arm) C 0.2 (thigh C leg)].
Functional ability test Handgrip | Change from baseline to after 40 minutes of continous cycling.
  Handgrip dynamometer was used for the upper body muscle strength evaluation. Both hands was tested.
Functional ability test 2-minute walk | Change from baseline to after 40 minutes of continous cycling.
  The two-minute walk test was applied where all the patients had to cover as far a distance as possible over 2 minutes. All the walking tests are related with the ability to perform independently the activities of daily living
Functional ability test 25-Foot Walk (T25-FW) | Change from baseline to after 40 minutes of continous cycling.
  The 25-Foot Walk (T25-FW) was used to measure the walking speed. It is a validated test that reflects the patient's mobility and leg function performance
Functional ability test five times sit-to-stand test (STS) | Change from baseline to after 40 minutes of continous cycling.
  The five times sit-to-stand test (STS) was used as an indicator for lower limb strength, balance and mobility. It has been reported that the STS times are associated with standing and leaning balance and mobility in older people. Slow STS time have been also found to predict subsequent disability, falls and hip fractures
Functional ability test Berg Balance Scale (BBS) | Change from baseline to after 40 minutes of continous cycling.
  The Berg Balance Scale (BBS) evaluates the performance in specific activities that require balance function. The BBS test lasts approximately 20 minutes and involves common actions (e.g. sit to stand, picking up an object, standing on one leg e.t.c.) necessary for activities of daily living. The BBS is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Functional ability test level of fatigue severity (FSS) | Change from baseline to after 40 minutes of continous cycling.
  The FSS is a 9-item self-report scale about fatigue of certain activities. Its score includes a 7-point scale from 1 = strongly disagree to 7 = strongly agree. The minimum possible score is nine and the highest is 63. High score indicates severe fatigue. FSS takes approximately eight minutes to complete.
Functional ability test Cognitive function | Change from baseline to after 40 minutes of continous cycling.
  Cognitive function was assessed with the mini mental state examination (MMSE) questionnaire. MMSE includes tests of orientation, attention, memory, language and visual-spatial skills. The answers in the MMSE are scored as following: 0=incorrect, 1=correct, 6= item administered, participant does not answer and 9= unknown
Functional ability test level of fatigue impact | Change from baseline to after 40 minutes of continous cycling.
  Level of fatigue was assessed by the Modified Fatigue Impact Scale (MFIS). The MFIS contains the following sections: a) Physical Sub-scale (score 0-36), b) Cognitive Sub-scale (score 0-40) and Psychological Sub-scale (score 0-8). The total MFIS score is 0-84; 0 represents the lower score and 84 represents the higher score.
Functional ability test level of fatigue inventory | Change from baseline to after 40 minutes of continous cycling.
  Level of fatigue was assessed by the 20-item scale Multidimensional Fatigue Inventory (MFI) questionnaire. The score of MFI is 1-7. The more the fatigue, the higher the score.
Functional ability test level of physical fatigue | Change from baseline to after 40 minutes of continous cycling.
  Level of fatigue was assessed by the Cognitive and Physical Fatigue in Multiple Sclerosis Scale (CPF-MS). The CPF-MS score is 1-5. The more the fatigue, the higher the score.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Kaltsatou, PhD, Principal Investigator — FAME Laboratory, Department of Exercise Science, University of Thessaly
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No